CLINICAL TRIAL: NCT00931359
Title: A Prospective, Multicenter, Parallel, Randomized, Blinded Study of the Efficacy and Safety of the DTS-G2 System in Patients With Axillary Hyperhidrosis
Brief Title: Efficacy and Safety of the DTS-G2 System in Patients With Axillary Hyperhidrosis
Acronym: DRI-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miramar Labs (Industry)
Responsible Party: Kathy O'Shaughnessy, VP Clinical/Regulatory, Miramar Labs, Inc
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CP-0003
Record Dates: First submitted 2009-06-28; First posted 2009-07-02 (Estimated); Results first posted 2011-06-14 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Primary Focal Hyperhidrosis, Axilla
Keywords: axillary; hyperhidrosis; primary focal
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment with DTS-G2 System (Experimental): Subjects receive treatment with the DTS-G2 System (an energy-based medical device) in both axilla. Multiple treatment sessions may be used.
  Interventions: Device: DTS-G2 System
- Sham treatment (Sham Comparator): All elements of the treatment are given except that no energy is delivered. Multiple treatment sessions may be used.
  Interventions: Device: DTS System (Sham treatment)

INTERVENTIONS:
Device: DTS-G2 System — Treatment with microwave energy
  Arms: Treatment with DTS-G2 System
Device: DTS System (Sham treatment) — Sham treatment - no energy is delivered
  Arms: Sham treatment

SUMMARY:
This is a prospective, multi-center, parallel, randomized, blinded study. The study has two groups, where in one study group the subjects receive treatment for axillary hyperhidrosis (excessive underarm sweating) with the DTS-G2 System in both axilla ("treatment group"). The other study group receives a sham treatment in both axilla where the subjects will have the same procedure performed but no energy from the device will be applied ("sham group"). Subjects will be randomized in a 2:1 ratio (treatment group: sham group).

Subjects enrolled in the study will be blinded regarding which study group they are in. The study hypothesis is that subjects that receive the treatment will have a reduction in underarm sweating compared to those in the sham group, as measured by a quality of life questionnaire.

All subjects will undergo follow up assessments at 14 days, 30 days, 3 months and 6 months post final treatment session. Subjects randomized to the treatment group will also have follow-up visits at 9 months and 12 months post final treatment session.

ELIGIBILITY:
Inclusion Criteria:

* baseline gravimetric measurement of spontaneous resting sweat production of at least 50 mg/5 min at room temperature in each axilla
* poor quality-of-life rating on the Hyperhidrosis Disease Severity Scale
* primary focal axillary hyperhidrosis evidenced by at least two of the standard criteria
* female subjects of child-bearing potential must not be pregnant or lactating and must agree to not become pregnant during the course of the study including follow-up period
* female subjects over 40 must have had a mammogram in the last 2 years
* subjects must be willing to comply with study visits and requirements

Exclusion Criteria:

* subject has secondary hyperhidrosis (e.g., endocrinopathy, medications)
* subject has active infection
* subject is pregnant or lactating
* subject has had prior surgery for axillary hyperhidrosis
* subject has had axillary injections of botulinum toxin A in the last year
* subject has used prescription antiperspirants in the last 14 days or plans to use them during the study period
* subject has used oral anticholinergics in the last 4 weeks
* subject is a prisoner or under incarceration
* subject is participating in a another clinical trial (or has in the last 30 days)
* subject has history of cancer (some exceptions)
* subject has a pacemaker or other electronic implant
* subject requires supplemental oxygen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dee Anna Glaser, MD, Principal Investigator — St. Louis University
Locations (7):
- United States (7):
  - Laser and Skin Surgery Center of Northern California, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - Bay Area Center for Plastic Surgery, Sunnyvale, California
  - The Coleman Clinic, Metairie, Louisiana
  - Skin Care Physicians, Chestnut Hill, Massachusetts
  - St Louis University, St Louis, Missouri
  - The Dermatology Group, Verona, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Treatment: Subjects received a sham treatment in two treatment sessions.
- Treatment With DTS-G2 System: Subjects received treatment in one to three treatment sessions with fixed device settings. Settings were at a generator output energy of 220J.
Period: Overall Study
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Started | 39 | 81
Completed | 33 | 68
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham Treatment | Treatment With DTS-G2 System | Total
Number analyzed (Participants) | 39 | 81 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 80 | 119
  >=65 years | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 34.1 (11.2) | 32.2 (10.7) | 32.8 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 44 | 70
  Male | 13 | 37 | 50
Region of Enrollment [Number; unit: participants]
  United States | 39 | 81 | 120

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects That Report an HDSS Score of 1 or 2 at 30 Days.
Description: The Hyperhidrosis Disease Severity Scale (HDSS) is a validated scale for measuring the effect of excessive sweating on the quality of life. It is a 4-point scale, with the following descriptors:
  1. - My underarm sweating is never noticeable and never interferes with my daily activities
  2. - My underarm sweating is tolerable but sometimes interferes with my daily activities
  3. - My underarm sweating is barely tolerable and frequently interferes with my daily activities
  4. - My underarm sweating is intolerable and always interferes with my daily activities
Time Frame: 30 days post-treatment
Population: Intent to Treat Population was used. Last Observation Carry Forward was used for missing data.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Number analyzed (Participants) | 39 | 81
Percentage of Participants | 54 | 89
Statistical Analysis 1: Comparison: Sham Treatment vs Treatment With DTS-G2 System; Test type: Superiority or Other; p < 0.001, ANOVA; Factors of treatment group and analysis center were considered

2. Secondary Outcome: Percentage of Subjects That Report an HDSS Score of 1 or 2 at the 6 Month Follow-up Visit.
Description: as for outcome 1
Time Frame: 6 months post-treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Number analyzed (Participants) | 39 | 81
Percentage of Participants | 44 | 67
Statistical Analysis 1: Comparison: Sham Treatment vs Treatment With DTS-G2 System; Test type: Superiority or Other; p = 0.019, ANOVA

3. Secondary Outcome: Percentage of Treatment Group Subjects That Report an HDSS Score of 1 or 2 at the 12 Month Visit
Description: The Hyperhidrosis Disease Severity Scale (HDSS) is a 4-point validated scale for measuring the effect of excessive sweating.
  1. - My underarm sweating is never noticeable and never interferes with my daily activities
  2. - My underarm sweating is tolerable but sometimes interferes with my daily activities
  3. - My underarm sweating is barely tolerable and frequently interferes with my daily activities
  4. - My underarm sweating is intolerable and always interferes with my daily activities This outcome is only measured for the treatment group; sham group exited the study after 6 month visit.
Time Frame: 12 months
Population: Sham group subjects exited the study after the 6 month follow-up visit, so were not in the study at this timepoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Number analyzed (Participants) | 0 | 81
Percentage of Participants |  | 69

4. Secondary Outcome: Percentage of Subjects With Reported Adverse Events
Description: Adverse events were defined in the protocol and included anticipated side effects of the procedure. These events were tracked by the clinical site and did include subject-reported events. The events reported here only included side effects that were attributed by the principal investigator as being possibly to definitely related to the device or procedure. They did not include expected treatment effects, such as swelling or bruising in the treatment area.
Time Frame: 6 months post-treatment
Measure: Number; unit: Percentage of Participants
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Number analyzed (Participants) | 39 | 81
Percentage of Participants | 13 | 28

ADVERSE EVENTS:
Time Frame: Sham group subjects followed for 6 months post-treatment. Treatment group subjects followed for 12 months post-treatment
Description: Only adverse events judged by investigator as being possibly, to definitely related to the device or procedure are listed.
Arm/Group | Sham Treatment | Treatment With DTS-G2 System
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/81
Other Adverse Events (participants affected / at risk) | 3/39 | 13/81
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham Treatment (N=39) | Treatment With DTS-G2 System (N=81)
Altered sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 8 (9)
Pain/soreness (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6)

LIMITATIONS AND CAVEATS:
Sham subjects exited the study at 6 months, so group comparisons are not possible for later timepoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days